CLINICAL TRIAL: NCT01103141
Title: Femoral Micropuncture or Routine Introducer Study
Acronym: FEMORIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This original design is no longer consistent with current clinical practice.
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 09-012
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Complications
Keywords: Vascular Surgical Procedures; Angioplasty; Radiology, Interventional

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Micropuncture (Active Comparator)
  Interventions: Device: Micropuncture needle set
- Standard (Active Comparator)
  Interventions: Device: Standard gauge-18 needle set

INTERVENTIONS:
Device: Micropuncture needle set — Groin access for vascular intervention
  Arms: Micropuncture
Device: Standard gauge-18 needle set — Groin access for vascular intervention
  Arms: Standard

SUMMARY:
FEMORIS is a marketing study approved by institutional review boards to compare the rates of complications found when using either the Micropuncture® needle introducer or a standard gauge-18 needle to access the groin blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing left heart catheterization with anticipated or possible percutaneous coronary intervention

Exclusion Criteria:

* Left heart cardiac catheterization purely for diagnostic purposes where percutaneous coronary intervention is not anticipated
* Catheterization utilizes primary vascular access site other than the groin
* Catheterization is intended for right heart procedure alone or combined with left and right heart procedures
* Age less than 18 years
* Patient has planned intervention or access utilizing the same groin within 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Francisco, Fresno, School of Medicine, Fresno, California
  - St. Vincent Hospital, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Micropuncture: Gauge-21 Micropuncture® needle
- Routine Access: Standard gauge-18 large-bore needle
Period: Overall Study
Arm/Group | Micropuncture | Routine Access
Started | 67 | 76
Completed | 65 | 74
Not Completed | 2 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micropuncture | Routine Access | Total
Number analyzed (Participants) | 67 | 76 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (11.3) | 63 (12.3) | 62.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 30 | 49
  Male | 48 | 46 | 94

OUTCOME MEASURES:

1. Primary Outcome: Major Peripheral Vascular Events
Description: Major peripheral vascular events occurring during femoral catheterization followed by Percutaneous Coronary Intervention (PCI), which include any of the following: Groin bleeding, including oozing or spurting after standard compression time necessitating further compression; Groin hematoma ≥ 5 cm at any time during or after the procedure; Pseudoaneurysm, confirmed by Doppler ultrasound; Arteriovenous (AV) fistula, confirmed by Doppler ultrasound; Arterial dissection, thrombosis, or embolism; Retroperitoneal bleeding defined by Computed Tomography Angiography (CTA) or surgery; Significant drop in hemoglobin ≥ 3 g/dL, or a drop in hematocrit ≥ 10% within 24-48 hours after the procedure compared to baseline without an obvious non-groin source; Any groin complication delaying hospital discharge; Large ecchymosis (> 15 cm) at the site of vascular access on follow-up (dark purple to black and confluent ecchymoses); Obvious extravascular extravasation of contrast as noted on the femoral
Time Frame: 7 - 14 days
Measure: Number; unit: participants
Arm/Group | Micropuncture | Routine Access
Number analyzed (Participants) | 67 | 76
participants
  Groin bleeding | 4 | 5
  Groin hematoma | 2 | 5
  Ecchymosis > 15 cm | 6 | 5

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | Micropuncture | Routine Access
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/76
Other Adverse Events (participants affected / at risk) | 12/67 | 15/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micropuncture (N=67) | Routine Access (N=76)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micropuncture (N=67) | Routine Access (N=76)
Ecchymosis > 15 cm (Injury, poisoning and procedural complications) | 6 (6) | 5 (5) — Ecchymosis > 15 cm at the vascular access site seen during follow-up
Groin bleeding (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) — Groin bleeding including oozing or spurting after standard compression time necessitating further compression
Groin hematoma (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) — Groin hematoma ≥ 5 cm noted at any time during or after the procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days